CLINICAL TRIAL: NCT03282227
Title: A Long-Term, Open-Label Study to Evaluate the Safety of M207 (Zolmitriptan Intracutaneous Microneedle System) in the Acute Treatment of Migraine
Brief Title: A Study to Evaluate the Long-Term Safety of M207 in the Acute Treatment of Migraine
Acronym: ADAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zosano Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-2017-001
Record Dates: First submitted 2017-09-05; First posted 2017-09-13 (Actual); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Migraine
Keywords: migraine; migraine headache; acute migraine; acute migraine headache
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Single dose, open-label treatment
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- M207 Microneedle System 3.8 mg (Experimental): M207 Microneedle System 3.8 mg (1.9 mg/patch x 2 patches)
  Interventions: Drug: M207 Microneedle System

INTERVENTIONS:
Drug: M207 Microneedle System — M207 Microneedle System 3.8 mg
  Other Names: ZP-Zolmitriptan Intracutaneous Microneedle System; ADAM-Zolmitriptan

SUMMARY:
This is an open-label, twelve-month safety study. There is a screening period followed by a run-in period to record migraine activity. Qualified subjects will receive study medication for up to twelve months for the treatment of multiple migraine attacks. Using the electronic diary (eDiary) to confirm they are experiencing a qualified migraine, subjects will self-administer the patches and respond to questions in the eDiary post treatment administration.

DETAILED DESCRIPTION:
This is an open-label, twelve-month safety study. There is a screening period followed by a run-in period (14 to 21 days) to determine eligibility for treatment with study medication based on daily eDiary data collection. Qualified subjects will receive study medication on Day 1 for up to twelve months for the treatment of migraine headaches. Migraines will be treated with a single dose, consisting of two patches, but subjects can treat multiple migraine attacks throughout the 12 months. Using the eDiary to confirm they are experiencing a qualified migraine, subjects will self-administer the patches and continue to respond to questions in the eDiary for 48 hours post treatment administration.

ELIGIBILITY:
Main Inclusion Criteria:

1. Women or men 18 to 75 years of age
2. Greater than 1 year history of episodic, migraine (with or without aura) with onset prior to 50 years of age.
3. Migraine history during the prior 6 months must include:

   1. at least 2 migraines per month
   2. no more than 8 migraines per month
   3. no more than 15 headache days per month
4. Women of child-bearing potential must not be pregnant, must agree to avoid pregnancy and use an acceptable double-barrier method of birth control during the trial.
5. Willing and able to treat a minimum of 2 migraines per month with study medication and consistently complete eDiary for up to 12 months.

Main Exclusion Criteria:

1. Contraindication to triptans
2. Use of selective serotonin reuptake inhibitors (drugs like Prozac®) or serotonin or norepinephrine reuptake inhibitors (drugs like Effexor®) or anti-coagulants (drugs like Coumadin®)
3. Known allergy or sensitivity to zolmitriptan or its derivatives or formulations
4. Known allergy or sensitivity to adhesives and/or titanium
5. Women who are pregnant, breast-feeding or plan a pregnancy during this study
6. Three or more of the following cardiovascular risk factors:

   * Current tobacco use
   * Hypertension or receiving anti-hypertensive medication for hypertension
   * Hyperlipidemia or on prescribed anti-cholesterol treatment
   * Family history of premature coronary artery disease
   * Diabetes mellitus
7. History or current abuse or dependence on alcohol or drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Kellerman, Pharm.D., Study Director — Zosano Pharma Corporation
Locations (31):
- United States (31):
  - Achieve Clinical Research, Birmingham, Alabama
  - Elite Clinical Studies, Phoenix, Arizona
  - Downtown L.A. Research Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Allergy Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Empire Clinical Research, Upland, California
  - Colorado Allergy Asthma Centers, Denver, Colorado
  - Harmony Medical Research Institute, Hialeah, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - DelRicht Research, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Michigan Headache and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research Institute, Plymouth, Minnesota
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Clinvest Research, Springfield, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Rochester Clinical Research, Rochester, New York
  - Peters Medical Research, High Point, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Raleigh Medical Group PMG Research, Raleigh, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Primary Care Associates/Radiant Research, Anderson, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - University of Texas Southwestern Medical Center - Neurology Clinic, Dallas, Texas
  - Central Texas Health Research, New Braunfels, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nahas SJ, Hindiyeh N, Friedman DI, Elbuluk N, Kellerman DJ, Foreman PK, Schmidt P. Long term safety, tolerability, and efficacy of intracutaneous zolmitriptan (M207) in the acute treatment of migraine. J Headache Pain. 2021 May 17;22(1):37. doi: 10.1186/s10194-021-01249-z. PMID 34001002

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | M207 Microneedle System 3.8 mg
Started | 342
Completed at Least 6 Months | 257
Completed (Completed 12 Months) | 127
Not Completed | 215
Not completed — Exposure Goals Achieved | 60
Not completed — Non-compliance w/ protocol requirements | 79
Not completed — Adverse Event | 15
Not completed — Lost to Follow-up | 21
Not completed — Withdrawal by Subject | 20
Not completed — Lack of Efficacy | 12
Not completed — Sponsor decision | 3
Not completed — Physician Decision | 2
Not completed — Pregnancy | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Safety population included 335 subjects (98.0%) who received any amount of study drug (applied at least 1 patch).
Arm/Group | M207 Microneedle System 3.8 mg
Number analyzed (Participants) | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 297
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60
  Not Hispanic or Latino | 275
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 55
  White | 265
  More than one race | 4
  Unknown or Not Reported | 3
Height [Mean (Standard Deviation); unit: cm] | 165.20 (8.602)
Weight [Mean (Standard Deviation); unit: kg] | 79.76 (20.847)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.19 (7.185)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Treatment-emergent Adverse Events (TEAE) Over 12 Months
Description: Number and % of subjects in safety population with any treatment-emergent adverse event(s) during the study. TEAE is defined as any new adverse event (AE) that started after first patch application. This was an open-label study with no control group. No statistical analyses were performed. Application site skin reactions including erythema, swelling, haemorrhage, bruise, pain, and pruritus were collected systematically via subject e-diary and/or investigator skin assessment at study visits. All other AEs were spontaneously reported by subject or observed upon examination.
Time Frame: 0 to 12 months
Population: Safety Population included 335 subjects (98.0%) who received any amount of study drug (applied at least 1 patch).
Measure: Count of Participants; unit: Participants
Arm/Group | M207 Microneedle System 3.8 mg
Number analyzed (Participants) | 335
Participants | 323

2. Secondary Outcome: Percentage of Migraine Attacks for Which Pain Freedom Was Achieved at 2 Hours Post-dose
Description: Percentage of migraine attacks for which pain freedom defined as a pain level of 'None' (Grade 0 on pain severity scale where 0: None, 1: Mild, 2: Moderate, 3: Severe, and lower values represent a better outcome) was achieved at 2 hours post-dose without the use of rescue medication. This was an open-label study with no control group. No statistical analyses were performed.
Time Frame: 2 hours for each Migraine, up to 12 months for each subject
Population: Modified intent-to-treat (mITT) Population included all subjects who received any amount of study drug to treat a qualifying migraine, and who had efficacy data.
Measure: Count of Units; unit: Qualifying migraines with 2 hour data
Units Other Than Participants: Qualifying migraines with 2 hour data
Arm/Group | M207 Microneedle System 3.8 mg
Number analyzed (Participants) | 335
Number analyzed (Qualifying migraines with 2 hour data) | 5617
Qualifying migraines with 2 hour data | 2477

3. Secondary Outcome: Percentage of Migraine Attacks for Which Most Bothersome Symptom Freedom Was Achieved at 2 Hours Post-dose
Description: Percentage of migraine attacks for which freedom from most bothersome symptom other than pain defined as an absence of the most bothersome symptom was achieved at 2 hours post-dose without the use of rescue medication. This was an open-label study with no control group. No statistical analyses were performed.
Time Frame: 2 hours for each Migraine, up to 12 months for each subject
Population: Modified Intent-to-Treat Population included all subjects who received
Measure: Count of Units; unit: Qualifying migraines with 2 hr data
Units Other Than Participants: Qualifying migraines with 2 hr data
Arm/Group | M207 Microneedle System 3.8 mg
Number analyzed (Participants) | 335
Number analyzed (Qualifying migraines with 2 hr data) | 5330
Qualifying migraines with 2 hr data | 3315

4. Secondary Outcome: Percentage of Migraine Attacks for Which Pain Relief Was Achieved at 2 Hours Post-dose
Description: Percentage of migraine attacks for which pain relief defined as an improvement of pain severity (1) to mild (Grade 1) or none (Grade 0) from moderate (Grade 2) or severe (Grade 3) at baseline, or (2) an improvement of pain severity to none (Grade 0) from mild (Grade 1) at baseline, without rescue medication was achieved. Pain severity scale has grades: 0: None, 1: Mild, 2: Moderate, 3: Severe, where lower values represent a better outcome. This was an open-label study with no control group. No statistical analyses were performed.
Time Frame: 2 hours for each Migraine, up to 12 months for each subject
Population: as for outcome 2
Measure: Count of Units; unit: Qualifying migraines with 2 hr data
Units Other Than Participants: Qualifying migraines with 2 hr data
Arm/Group | M207 Microneedle System 3.8 mg
Number analyzed (Participants) | 335
Number analyzed (Qualifying migraines with 2 hr data) | 5617
Qualifying migraines with 2 hr data | 4552

5. Secondary Outcome: Percentage of Migraine Attacks for Which Nausea Freedom Was Achieved at 2 Hours Post-dose
Description: Percentage of subjects for which nausea freedom defined as absence of nausea and/or vomiting without the use of rescue medication was achieved at 2 hours post-dose. This was an open-label study with no control group. No statistical analyses were performed.
Time Frame: 2 hours for each Migraine, up to 12 months for each subject
Population: as for outcome 2
Measure: Count of Units; unit: Qualifying migraines with 2 hr data
Units Other Than Participants: Qualifying migraines with 2 hr data
Arm/Group | M207 Microneedle System 3.8 mg
Number analyzed (Participants) | 335
Number analyzed (Qualifying migraines with 2 hr data) | 5617
Qualifying migraines with 2 hr data | 4628

6. Secondary Outcome: Percentage of Migraine Attacks for Which Photophobia Freedom Was Achieved at 2 Hours Post-dose
Description: Percentage of migraine attacks for which photophobia freedom defined as an absence of photophobia without the use of rescue medication was achieved at 2 hours post-dose. This was an open-label study with no control group. No statistical analyses were performed.
Time Frame: 2 hours for each Migraine, up to 12 months for each subject
Population: as for outcome 2
Measure: Count of Units; unit: Qualifying migraines with 2 hour data
Units Other Than Participants: Qualifying migraines with 2 hour data
Arm/Group | M207 Microneedle System 3.8 mg
Number analyzed (Participants) | 335
Number analyzed (Qualifying migraines with 2 hour data) | 5617
Qualifying migraines with 2 hour data | 3410

7. Secondary Outcome: Percentage of Migraine Attacks for Which Phonophobia Freedom Was Achieved at 2 Hours Post-dose
Description: Percentage of migraine attacks for which phonophobia freedom defined as an absence of phonophobia without the use of rescue medication was achieved at 2 hours post-dose. This was an open-label study with no control group. No statistical analyses were performed.
Time Frame: 2 hours for each Migraine, up to 12 months for each subject
Population: as for outcome 2
Measure: Count of Units; unit: Qualifying migraines with 2 hour data
Units Other Than Participants: Qualifying migraines with 2 hour data
Arm/Group | M207 Microneedle System 3.8 mg
Number analyzed (Participants) | 335
Number analyzed (Qualifying migraines with 2 hour data) | 5617
Qualifying migraines with 2 hour data | 3563

ADVERSE EVENTS:
Time Frame: 0-12 months
Description: Application site skin reactions including erythema, swelling, haemorrhage, bruise, pain, and pruritus were collected systematically via subject e-diary and/or investigator skin assessment at study visits. All other AEs were spontaneously reported by subject or observed upon examination.
Arm/Group | M207 Microneedle System 3.8 mg
All-Cause Mortality (participants affected / at risk) | 0/335
Serious Adverse Events (participants affected / at risk) | 5/335
Other Adverse Events (participants affected / at risk) | 323/335
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | M207 Microneedle System 3.8 mg (N=335)
Hypokalaemia (Metabolism and nutrition disorders) | 1
Foetal disorder (Congenital, familial and genetic disorders) | 1 — Fetal chromosomal disorder
Procedural pain (Nervous system disorders) | 1
Breast cancer stage II (Reproductive system and breast disorders) | 1
Pneumonia (Infections and infestations) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | M207 Microneedle System 3.8 mg (N=335)
Application site erythema (Skin and subcutaneous tissue disorders) | 316
Application site swelling (Skin and subcutaneous tissue disorders) | 296
Application site haemorrhage (Skin and subcutaneous tissue disorders) | 225
Application site bruise (Skin and subcutaneous tissue disorders) | 194
Application site pain (Skin and subcutaneous tissue disorders) | 81
Application site discolouration (Skin and subcutaneous tissue disorders) | 53
Application site pruritus (Skin and subcutaneous tissue disorders) | 52
Application site oedema (Skin and subcutaneous tissue disorders) | 8
Upper respiratory tract infection (Infections and infestations) | 28
Sinusitis (Infections and infestations) | 13
Viral upper respiratory tract infection (Infections and infestations) | 7
Nausea (Gastrointestinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT03282227/SAP_000.pdf
  • Study Protocol (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03282227/Prot_001.pdf